CLINICAL TRIAL: NCT02162589
Title: Peroral Endoscopic Myotomy (POEM) For The Treatment Of Achalasia: A Retrospective And Prospective Multicenter Registry.
Brief Title: Peroral Endoscopic Myotomy (POEM) For The Treatment Of Achalasia: A Registry
Acronym: POEM Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Michel Kahaleh, Chief of Endoscopy, Weill Medical College of Cornell University
Other Study IDs: 1309014292
Record Dates: First submitted 2014-06-10; First posted 2014-06-12 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Achalasia
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- POEM for Achalasia: Any patient who has undergone clinically indicated and/or standard of care POEM for the treatment of Achalasia.
  Interventions: Procedure: POEM

INTERVENTIONS:
Procedure: POEM — Per oral endoscopic myotomy

SUMMARY:
Prospective Multicenter registry study to assess the safety and efficacy of clinically indicated peroral endoscopic myotomy (POEM) for the treatment of Achalasia

DETAILED DESCRIPTION:
Our institution performs therapeutic Interventional Endoscopy in around 700-1000 patients a year. We come across several patients with esophageal disorders, including esophageal cancer and Achalasia.

Achalasia is an uncommon esophageal motility disorder caused by the inability of the lower esophageal sphincter (LES) to relax due to the degeneration of inhibitory neurons in the myenteric plexus. (1,2) Evidence of achalasia in patients includes the absence of relaxation in the LES, abnormal swallowing relaxation of the LES, or the absence of peristalsis in the esophageal body.

(2,3 ) Treatments for achalasia primarily focus on forcing the relaxation of the LES. Conventional treatments such as botolinum toxin (Botox) injections, balloon dilation, nitrate and calcium antagonists, and Heller myotomy, although effective, have many disadvantages. (4,5, 6) Balloon dilation, which is the least noninvasive out of the non-surgical processes, can still result in esophageal perforation and its long term investigations have reported unfavorable (2). Surgical myotomies, such as Heller myotomy and laproscopic esophagomytomy, are indicated when non-surgical therapies render ineffective.

However, gastroesophageal reflux disease occurs in 30% (7) of Heller Myotomy patients and it has a 10-15% failure rate (8). Per-oral endoscopic myotomy (POEM), derived from Advances in Natural Orifice Transluminal Endoscopic Surgery (NOTES) and advances in submucosal dissection (9,10,11), presents a novel, less invasive, and permanent treatment to lower esophageal sphincter pressure (12). POEM was first described by Parischa et al in porcine models in 2007 and its introduction into clinical care in 17 patients was made by Inoue et al in 2010. (12,13) POEM is performed entirely endoscopically, enabling much deeper incisions in the thoracic esophagus than surgery is able to create. (2 , 13) An incision is made in the mid- esophagus by creating a submucosal tunnel to access the muscle layer all the way down to the gastric cardia and conduct myotomy (partial muscle removal). Partial inner circular muscle layer is removed from the last part of the esophagus, lower esophageal sphincter and the upper part of the stomach. After the myotomy is completed, endoclips are used to seal the incision and the endoscope is withdrawn. (2) The effectiveness of POEM is indicated by patient studies based mostly in Europe and Asia. Recent studies report POEM has a 90% effectiveness rate compared to patients who have undergone Heller myotomy. (9 ,14,15) Based on study design and results of the recent studies done in Europe and Asia (retrospective only), we would like to evaluate and verify technical feasibility, clinical success and safety of clinically indicated POEM for Achalasia prospectively with a longer follow up duration (more than 6 months). Evaluation of these factors would help us compare them to conventional treatment modalities within our current facility; and consequently help us identify appropriate treatment techniques and improve clinical management of patients at WCMC-NYPH. The purpose of this retrospective and prospective registry is to assess long term data on efficacy, safety and clinical outcome of POEM. The registry will evaluate technical feasibility, clinical outcome, safety profile and overall clinical management through medical chart review.

The procedures we are evaluating are all clinically indicated and will not be prescribed to someone to participate in this registry study.

The purpose of this retrospective and prospective registry is to assess long term data on efficacy, safety and clinical outcome of POEM. The registry will evaluate technical feasibility, clinical outcome, safety profile and overall clinical management through medical chart review.

Study Design: Retrospective and Prospective, observational, medical chart review for at least 6 standard of care visits up to 1 year after subject consents for study participation.

Interventions: None Subject Participation: Subject's participation in this study will allow us to collect data for at least 6 standard of care visits up to 1 year after consenting to participating in this registry study. Subject will undergo a standard of care or clinically indicated Endoscopic procedure and POEM and subsequent follow up clinic visits as part of their standard medical care.

Subject will sign a separate clinical consent for the Endoscopic procedure and placement of the sutures(s). That consent form will explain the procedure as well as the risks involved with the procedure. Subject will undergo endoscopic procedures and POEM and subsequent follow up clinic visits regardless of their participation in this study. Subject will undergo no additional tests and procedures as part of this study.

Study duration: At least 6 standard of care visits up to 1 year for each subject . Once the subject consents, data will be collected for their clinically indicated or standard of care procedure visit and follow up visits.

Research related activities: Consenting, medical chart review and case report form entry.

Clinically indicated and necessary procedures include: Evaluation, imaging, lab tests, adverse events monitoring and POEM.

Standard of care follow up visits for POEM are usually 15 days, 1 month, 3 months, 6 months and 12 months post procedure. All data will be collected from Medical charts. No subject surveys or questionnaires will be administered.

Study Design at Coordinating Center - Primary site (WCMC): T All patients who have had clinically indicated POEM done for Achalasia.

Study Design at Secondary site: Other sites must have either a database review protocol and/or a clinical trial that would collect data on POEM prior to participating in the registry.

These sites would have IRB approved protocols to collect and send procedure data to the primary site (WCMC). Additionally, the secondary study sites would mention WCMC as an entity that could receive PHI in their respective protocols and consent/HIPAA forms. All secondary study sites' IRB approvals will be sent to the primary/coordinating study center for WCMC IRB.

Data sharing agreements will be finalized prior to sharing of any and all confidential data.

Registry Hosting: The coordinating center and primary site (WCMC) will host the registry on the local servers. Electronic Data Capture (EDC) system REDCAP will be used for data entry, compilation and querying. Secondary sites will be trained and a Redcap login ID will be provided. REDCAP data from all sites will be accessible only to the primary coordinating site investigators. The data will be stored on the REDCAP server. Specific access/editing permissions will be granted as per standard protocol to personnel at secondary sites who will enter data.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient who has undergone clinically indicated and/or standard of care POEM for the treatment of Achalasia
2. Above or equal to 18 years of age

Exclusion Criteria:

1. Any patient who has not undergone POEM for the treatment of Achalasia
2. Below 18 years of age

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient who has undergone clinically indicated and/or standard of care POEM for the treatment of Achalasia and above or equal to 18 years of age
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-02; Primary Completion 2017-12-01 (Estimated); Study Completion 2018-01-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Success | 1 year
  Documentation of clinical success rates such as achievement of symptoms remission (dysphagia, reflux, etc.) and reduced lower esophageal sphincter pressures (manometry).

SECONDARY OUTCOMES:
Safety Rate | 6 months
  Documentation of Safety: Number of subjects with Adverse Events, Type, frequency and intensity of adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No IPD sharing

REFERENCES:
- [Background] Kumta NA, Mehta S, Kedia P, Weaver K, Sharaiha RZ, Fukami N, Minami H, Casas F, Gaidhane M, Lambroza A, Kahaleh M. Peroral endoscopic myotomy: establishing a new program. Clin Endosc. 2014 Sep;47(5):389-97. doi: 10.5946/ce.2014.47.5.389. Epub 2014 Sep 30. PMID 25324996
- [Derived] Tyberg A, Seewald S, Sharaiha RZ, Martinez G, Desai AP, Kumta NA, Lambroza A, Sethi A, Reavis KM, DeRoche K, Gaidhane M, Talbot M, Saxena P, Zamarripa F, Barret M, Eleftheriadis N, Balassone V, Inoue H, Kahaleh M. A multicenter international registry of redo per-oral endoscopic myotomy (POEM) after failed POEM. Gastrointest Endosc. 2017 Jun;85(6):1208-1211. doi: 10.1016/j.gie.2016.10.015. Epub 2016 Oct 15. PMID 27756611
- See also: Description of POEM procedure for Achalasia — http://www.youtube.com/watch?v=oWp3pjhaJWo